CLINICAL TRIAL: NCT05495191
Title: Association Between Signal Intensity Gradient of Cerebral Arteries From Time-of-flight Magnetic Resonance Angiography and Clinical Outcome in Patients With Lenticulostriate Artery Infarction
Brief Title: Signal Intensity Gradient in Cerebral Arteries
Status: Completed | Type: Observational
Sponsor: Chonbuk National University Hospital (Other)
Collaborators: Korean Society of Neurosonology (Unknown); Ministry of SMEs and Startups, Republic of Korea (Unknown); Korean Neurological Association (Unknown)
Responsible Party: Sponsor
Other Study IDs: SIGLSA
Record Dates: First submitted 2022-08-03; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Ischemic Stroke, Acute
Keywords: Cerebral artery; Lenticulostriate artery infarction; Signal intensity gradient; Signal intensity gradient, Wall shear stress
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grouped as the favorable outcome: <3 mRS of discharge or 7th day in the patients with the lenticulostriate artery infarction
  Interventions: Diagnostic Test: Signal intensity gradient
- Grouped as the unfavorable outcome: ≥3 mRS of discharge or 7th day in the patients with the lenticulostriate artery infarction
  Interventions: Diagnostic Test: Signal intensity gradient

INTERVENTIONS:
Diagnostic Test: Signal intensity gradient — In time-of-flight (TOF) MRA, The signal intensities at the iso-point (Φa; signal intensity at position A [Xa] along the arterial contour line) and at the inner point (Φb; signal intensity at position B [Xb]) were calculated by using a trilinear interpolation algorithm based on the positions and signal intensities in the eight neighboring voxels. The signal intensities of TOF-MRA were normalized to eliminate the offset and scale effects across the MRA datasets of participants. For each iso-point (position A), the SIG was calculated from the difference in signal intensities between points A and B as follows:
  Scalar SIG, SI/mm = (Φb - Φa) / │Xb - Xa│ (1)
  Vector SIG, SI/mm = (Φb - Φa) n / │Xb - Xa│ (2)

SUMMARY:
Arterial wall shear stress (WSS) contributes to atherosclerosis from its inception, progression, and disruption of plaque. However, there is no previous study for an association between cerebral artery WSS and clinical outcome in patients with ischemic stroke in lenticulostriate artery.

The researchers aimed to investigate whether the signal intensity gradient (SIG) from Time-of-Flight Magnetic Resonance Angiography (TOF MRA) in cerebral arteries, as a surrogate measure of arterial WSS, is associated with clinical outcome, which was determined with modified Rankin Scale (mRS).

The patients (n=294) with the lenticulostriate artery infarction were collected in 3 hospitals with variable locations and sizes (Gunsan, Jeonju, and Seoul). For a clinical outcome, National Institute of Health Stroke Scale (NIHSS) and modified Rankin Scale (mRS) were checked serially from the date of admission. The mRS 2 or less at the 7th day or discharge was defined as a favorable outcome. The arterial SIGs were measured concurrently in both internal carotid, anterior/middle/posterior cerebral, vertebral arteries, and basilar artery from TOF MRA on initial diagnosis. The independent association between the clinical outcome and cerebral arterial SIG was analyzed adjusting for all the possible potential confounders.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 years or older who had brain magnetic resonance imaging (MRI) for acute ischemic stroke within 3 days
2. Patients who underwent diffusion-weighted imaging (DWI) and apparent diffusion coefficient of the cerebral parenchyma, and cerebral angiographic measurements, in which, intracranial arteries should be examined by time-of-flight (TOF) techniques
3. A patient with high signal intensity lesions in the unilateral LSA territory on DWI.

Exclusion Criteria:

1. Patients younger than 18 years of age
2. Patients with moderate to severe (>50%) stenosis or occlusion of the major intracranial and extracranial arteries, including internal carotid artery (ICA), middle cerebral artery (MCA), anterior cerebral artery (ACA), posterior cerebral artery (PCA), basilar artery (BA), and vertebral artery (VA)
3. Patients whose ischemic stroke was due to or related with cardiac or rare etiology (e.g., arterial dissection, moyamoya disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a multi-center, retrospective cohort study for all consecutive patients. From January 2015 to March 2021, patients who were diagnosed with acute ischemic stroke in the lenticulostriate artery (LSA) territory were registered at three centers (Jeonbuk National University Hospital, Samsung Medical Center, and Gunsan Medical Center). The 3 centers have their own characteristics: Gunsan Medical center is in a small city where about 300,000 citizens live, Jeonbuk National University Hospital is in a medium sized city where about 650,000 citizens live, and Samsung Medical Center is in a capital city where about 10,000,000 citizens live).
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-07-23 (Actual)

PRIMARY OUTCOMES:
Change of signal intensity gradient at discharge or 7th day in the patients with the lenticulostriate artery infarction | Approximately 1 week
  Degrees of the signal intensity gradient (SIG) from brain TOF-MRA in major cerebral arteries are measured in the patients with the lenticulostriate artery infarction at discharge or 7th day.

CONTACTS AND LOCATIONS:
Overall Officials: Chan-Hyuk Lee, Dr., Principal Investigator — Jeonbuk National University Hospital
Locations (1):
- Jeonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Decavel P, Vuillier F, Moulin T. Lenticulostriate infarction. Front Neurol Neurosci. 2012;30:115-9. doi: 10.1159/000333606. Epub 2012 Feb 14. PMID 22377876
- [Background] Jeong SK, Lee JY, Rosenson RS. Association between Ischemic Stroke and Vascular Shear Stress in the Carotid Artery. J Clin Neurol. 2014 Apr;10(2):133-9. doi: 10.3988/jcn.2014.10.2.133. Epub 2014 Apr 23. PMID 24829599
- [Background] Han KS, Lee SH, Ryu HU, Park SH, Chung GH, Cho YI, Jeong SK. Direct Assessment of Wall Shear Stress by Signal Intensity Gradient from Time-of-Flight Magnetic Resonance Angiography. Biomed Res Int. 2017;2017:7087086. doi: 10.1155/2017/7087086. Epub 2017 Aug 16. PMID 28900625

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/91/NCT05495191/Prot_SAP_000.pdf